CLINICAL TRIAL: NCT00249613
Title: Gender-Responsive Treatment for Women Offenders
Brief Title: Gender-Responsive Treatment for Women Offenders - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael Prendergast, Research Historian, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-16277-1; R01DA016277 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-03

CONDITIONS: Substance Abuse Problem
Keywords: gender-responsive substance abuse treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Women-Only (Experimental): Substance abuse treatment program for women only
  Interventions: Behavioral: Women-Only
- Mixed-Gender (No Intervention): Substance abuse treatment program for both women and men

INTERVENTIONS:
Behavioral: Women-Only — Gender-responsive treatment for women only
  Arms: Women-Only

SUMMARY:
The purpose of this study is to determine whether substance abuse treatment designed specifically for drug-dependent women offenders provides better outcomes than standard drug court treatment (mixed-gender programs).

DETAILED DESCRIPTION:
In this five-year study, a total of 300 women entering court-referred treatment throughout Los Angeles County and who agree to participate in the study will be randomly assigned to a women-focused or to a mixed-gender outpatient treatment program. The study will assess the impact of women-focused substance abuse treatment using outcome measures including recidivism, substance abuse and relapse, and social adjustment (e.g., employment, parenting behaviors, psychological improvement, and HIV risk reduction behaviors), compared to the impact of traditional mixed-gender programs. Assessments will occur at baseline and at 1 month, 12 months, and 24 months after admission.

ELIGIBILITY:
Inclusion Criteria:

* Drug court participant
* At least eighteen (18) years old
* Have had no more than three prior non-violent, non-drug felony convictions
* Do not have a current charge of driving under the influence of alcohol or drugs or a charge of sale or transportation of drugs

Exclusion Criteria:

* Not capable of giving informed consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2005-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Prendergast, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California - Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Result] Prendergast ML, Messina NP, Hall EA, Warda US. The relative effectiveness of women-only and mixed-gender treatment for substance-abusing women. J Subst Abuse Treat. 2011 Jun;40(4):336-48. doi: 10.1016/j.jsat.2010.12.001. Epub 2011 Feb 11. PMID 21315540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 425 Potential subjects approached at community drug treatment clinics and drug courts 291 Completed baseline intake interview
Pre-assignment Details: At baseline, we had 51 Refusals, 30 Ineligible for study 27 No show to baseline interview, and 26 who did not complete baseline intake interview.
Groups:
- Women-Only Treatment 152 Subjects: Out patient gender-responsive substance abuse treatment for women only
- Mixed-Gender Treatment 139 Subjects: Out-patient substance abuse treatment that included both women and men
Period: Baseline
Arm/Group | Women-Only Treatment 152 Subjects | Mixed-Gender Treatment 139 Subjects
Started | 152 | 139
Completed | 152 | 139
Not Completed | 0 | 0
Period: 12 Month Follow-up
Arm/Group | Women-Only Treatment 152 Subjects | Mixed-Gender Treatment 139 Subjects
Started | 152 | 139
Completed | 135 | 124
Not Completed | 17 | 15
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Women-Only Treatment 152 Subjects: Out-patient gender-responsive substance abuse treatment for women only
- Mixed-Gender Treatment 139 Subjects: Out-patient substance abuse treatment for women and men
- Total: Total of all reporting groups
Arm/Group | Women-Only Treatment 152 Subjects | Mixed-Gender Treatment 139 Subjects | Total
Number analyzed (Participants) | 152 | 139 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (10.1) | 36.5 (10.2) | 35.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 139 | 291
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 152 | 139 | 291

OUTCOME MEASURES:

1. Primary Outcome: Results (Unadjusted) for Criminal Activities in Past 30 Days at Baseline and Follow-up for Women in Women-Only Treatment and Mixed-Gender Treatment
Time Frame: baseline and 1-year follow-up
Population: Intention to treat (ITT)
Measure: Number; unit: Percentage reporting criminal activity
Arm/Group | Women-Only | Mixed-Gender
Number analyzed (Participants) | 152 | 139
Percentage reporting criminal activity
  Baseline | 63.9 | 76.9
  1 Year Follow-up | 22.3 | 39.7

2. Primary Outcome: Predictors of Criminal Activity at 12 Months Post Intake
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: Odds ratio
Groups:
- Women-Only Compared to Mixed-Gender: Outpatient gender-responsive substance abuse treatment for women only compared to outpatient substance abuse treatment for women and men
Arm/Group | Women-Only Compared to Mixed-Gender
Number analyzed (Participants) | 259
Odds ratio | 0.40 [0.21 to 0.79]
Statistical Analysis 1: Comparison: Women-Only Compared to Mixed-Gender; Logistic regression does not separate arms because group status (women-only vs mixed gender) is the dependent variable in our multinomial logistic regression. Because we were not able to randomly assign after all, we also included a propensity score, and additional variables (substance use in past 30 days at baseline, age, race/ethnicity, childhood sexual abuse history, previous treatment, criminal justice funding source, and primary drug) to adjust for the non-random sampling; Test type: Superiority or Other; p = 0.01, Regression, Logistic — Odds ratio is 0.40, confidence interval is 0.21-0.79; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.21 to 0.79], Standard Error of Mean 0.34 — The direction of the comparison would dictate that odds ratio of less than 1 would indicate Women-Only participants are less likely than Mixed-Gender participants to engage in criminal activities

3. Secondary Outcome: Predictors of Change in Employment at 12 Months Post Intake: Generalized Estimating Equation (GEE) Model
Description: Predictors of change in employment at 12 months post intake: GEE - comparison of Women-Only vs. Mixed-Gender treatment models
Time Frame: 12 month post intake
Measure: Number (95% Confidence Interval); unit: Beta coefficient
Groups:
- Group Status (Women-Only Compared to Mixed-Gender): Outpatient gender-responsive substance abuse treatment for women only vs. outpatient mixed-gender substance abuse treatment
Arm/Group | Group Status (Women-Only Compared to Mixed-Gender)
Number analyzed (Participants) | 291
Beta coefficient | -0.70 [-2.11 to 0.70]
Statistical Analysis 1: Comparison: Group Status (Women-Only Compared to Mixed-Gender); Generalized estimating equation (GEE) models do not separate arms: group status (women-only vs mixed-gender) is the dependent variable. Because we were not able to randomly assign, we also included a propensity score, and additional variables (education, race/ethnicity, marital status, income, history of sexual abuse, criminal justice funding source, had child, mental health symptoms, and a time in treatment by group interaction term) to adjust for the non-random sampling; Test type: Superiority or Other; p = 0.33, Generalized estimating equations (GEE); Beta coefficient = -0.70, 95% CI 2-sided [-2.11 to 0.70], Standard Error of Mean 0.72

4. Primary Outcome: Any Substance Use Past 30 Days
Description: Substance use in past 30 days at 12 months post intake
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: Odds ratio
Groups:
- Group Status (Women-Only Compared to Mixed-Gender: Comparison of outcome in Women-Only vs. Mixed-Gender treatment
Arm/Group | Group Status (Women-Only Compared to Mixed-Gender
Number analyzed (Participants) | 291
Odds ratio | 0.42 [0.22 to 0.82]
Statistical Analysis 1: Comparison: Group Status (Women-Only Compared to Mixed-Gender; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.01, Regression, Logistic; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.22 to 0.82], Standard Error of Mean .34 — The direction of the comparison would dictate that odds ratio of less than 1 would indicate Women-Only treatment participants are less likely than the Mixed-Gender group to use drugs or alcohol during the 30 days prior to the 12-Mo follow-up

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Women-Only: Outpatient gender-responsive substance abuse treatment for women only
- Mixed-Gender: Outpatient mixed-gender substance abuse treatment
Arm/Group | Women-Only | Mixed-Gender
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/139
Other Adverse Events (participants affected / at risk) | 0/152 | 0/139

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No